CLINICAL TRIAL: NCT01502254
Title: Patients' Knowledge and Understanding of Cancer Clinical Trials - a Randomised Study of Audio Recorded Information
Brief Title: Patients' Knowledge and Understanding of Cancer Clinical Trials - a Study of Audio Recorded Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mia Bergenmar, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: QuIC-3
Record Dates: First submitted 2011-12-22; First posted 2011-12-30 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Cancer
Keywords: Informed consent; Cancer clinical trials; Patient information; Knowledge; Questionnaire; Patient Eligible for a Phase II or III Cancer Clinical Trial; Scheduled Clinical Visit for Information About a Trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Copy of audio recording (Experimental): Patients receive a copy of the audio recorded information about the clinical trial directly after the clinical visit. This makes it possible to repeat the information before a decision is made to participate in the clinical trial or not.
  Interventions: Other: audio recorded information
- No copy of audio recording (No Intervention): Patients in the control arm receive no copy of the audio recording.

INTERVENTIONS:
Other: audio recorded information — Access to the audio recorded information about the clinical trial the patient was information about and asked to consider. A copy of the audio recording is given to the patients directly after the clinical visit.
  Arms: Copy of audio recording

SUMMARY:
The purpose of this study is to test if cancer patients who are informed about, and offered participation in a cancer clinical trial, are more knowledgeable about cancer clinical trials if they have access to an audio recording of their information visit.

ELIGIBILITY:
Inclusion Criteria:

* Informed in Swedish about a phase II or III clinical trial
* Signed a consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Patients' knowledge about clinical trials measured by the questionnaire Quality of Informed Consent | The questionnaire is sent to patients within a week after consenting to the trial.
  The questionnaire is sent to patients within a week after consenting to the trial. One reminder is sent to those not responding within two weeks.

SECONDARY OUTCOMES:
Patients' perceived understanding of clinical trials measured by the questionnaire Quality of Informed Consent | The questionnaire is sent to patients within a week after consenting to the trial.
  The questionnaire is sent to patients within a week after consenting to the trial. One reminder is sent to those not responding within two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mia Bergenmar, PhD, Principal Investigator — Department of Oncology, Karolinska University Hospital and Department of Oncology-Pathology, Karolinska Institutet, Stockholm, Sweden
Locations (1):
- Department of Oncology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Bergenmar M, Molin C, Wilking N, Brandberg Y. Knowledge and understanding among cancer patients consenting to participate in clinical trials. Eur J Cancer. 2008 Nov;44(17):2627-33. doi: 10.1016/j.ejca.2008.08.013. Epub 2008 Sep 23. PMID 18818068
- [Background] Bergenmar M, Johansson H, Wilking N. Levels of knowledge and perceived understanding among participants in cancer clinical trials - factors related to the informed consent procedure. Clin Trials. 2011 Feb;8(1):77-84. doi: 10.1177/1740774510384516. Epub 2010 Nov 25. PMID 21109583
- [Derived] Bergenmar M, Johansson H, Wilking N, Hatschek T, Brandberg Y. Audio-recorded information to patients considering participation in cancer clinical trials - a randomized study. Acta Oncol. 2014 Sep;53(9):1197-204. doi: 10.3109/0284186X.2014.921726. Epub 2014 Jun 9. PMID 24909376